CLINICAL TRIAL: NCT03399851
Title: Comparison of Amplatzer Amulet vs Watchman Device in Patients Undergoing Left Atrial Appendage Closure: the SWISS-APERO Randomized Clinical Trial
Brief Title: Comparison of Amplatzer Amulet and Watchman Device in Patients Undergoing Left Atrial Appendage Closure. (SWISS-APERO)
Acronym: SWISS-APERO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWISS-APERO
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Left Atrial Appendage Closure
MeSH Terms: interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amplatzer Amulet (Active Comparator): Left atrial appendage closure (LAAC) with Amplatzer Amulet implantation will be performed according to device specific instruction for use, based on both TEE guidance and angiography, femoral venous access and inter-atrial septum crossing.
  Interventions: Device: Amplatzer Amulet for left atrial appendage closure
- Watchman/FLX (Active Comparator): Left atrial appendage closure (LAAC) with Watchman/FLX implantation will be performed according to device specific instruction for use, based on both TEE guidance and angiography, femoral venous access and inter-atrial septum crossing.
  Interventions: Device: Watchman/FLX for left atrial appendage closure

INTERVENTIONS:
Device: Amplatzer Amulet for left atrial appendage closure — The closure of the left atrial appendage (LAAC) is performed percutaneously. Implantation of the Amplatzer Amulet will be performed according to device specific instruction for use, based on both TEE guidance and angiography, femoral venous access and inter-atrial septum crossing.
  Arms: Amplatzer Amulet
Device: Watchman/FLX for left atrial appendage closure — The closure of the left atrial appendage (LAAC) is performed percutaneously. Implantation of the Watchman/FLX will be performed according to device specific instruction for use, based on both TEE guidance and angiography, femoral venous access and inter-atrial septum crossing.
  Arms: Watchman/FLX

SUMMARY:
Left atrial appendage closure (LAAC) is an emerging therapeutic option in non-valvular atrial fibrillation (NVAF) patients with high thromboembolic and bleeding risks. In Europe the devices most frequently utilized for LAAC are Amplatzer Amulet (St. Jude Medical-Abbott) and Watchman (Boston Scientific) system. However there are currently no randomized controlled trials assessing the degree of LAA closure between the two devices. The main purpose of this trial is to evaluate the feasibility and the efficacy of the devices in terms of LAA complete occlusion with a non-invasive imaging technique such as cardiac computed tomography angiography (CCTA).

DETAILED DESCRIPTION:
Non-valvular Atrial fibrillation (NVAF) is the most common cardiac arrhythmia and a major cause of morbidity and mortality because of cardioembolic stroke. Oral anticoagulation (OAC) with vitamin K antagonists (VKA) or Non-vitamin K antagonist anticoagulant (NOAC) is the most effective prophylaxis for stroke in NVAF. However (N)OAC therapy is associated with a significant bleeding liability and long-term (N)OAC therapy in patients with NVAF and concomitant high bleeding risk poses safety issues in a sizable and growing population in clinical practice. Thus, a new and emerging therapeutic option in this high-risk patient population is the left atrial appendage closure (LAAC). There are many available systems approved for percutaneous LAAC. One of the most widely used is the Watchman™ system (Boston Scientific), which was tested in the setting of two randomized control trials (RCT), which demonstrated the safety of the procedure and the non-inferiority in terms of stroke reduction compared to OAC. Another device largely used is the Amplatzer Amulet (St. Jude Medical-Abbott). There is no RCT comparing this device with OAC, but many prospective and retrospective studies had shown the same safety profile and the non-inferiority with the OAC. From the very beginning of the LAAC, a crucial assessment is the degree of LAA occlusion granted by the implanted device. Many imaging modalities have been used to assess LAA occlusion, including transesophageal echocardiography (TEE), fluoroscopy or cardiac computed tomography angiography (CCTA). In the setting of available randomized trials, successful closure was defined with the presence of a regurgitant flow ≤ 5 mm assessed with TEE. In the last years several groups assessed the value of CCTA as non-invasive post-procedural surveillance imaging modality after endovascular LAAC to evaluate atrial-side device thrombus, residual leak (and mechanisms thereof), device position, pericardial effusion and most importantly LAA patency. There are currently no randomized controlled trials assessing the degree of LAA occlusion between Amulet and Watchman.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female subject aged 18 years or more with no upper age limit and willing to comply with the protocol
* Indication to a LAAC as indicated in study population (HAS BLEED ≥3 or High bleeding risk as defined by Munich consensus document and CHA2DS2-VASc≥2)

Exclusion Criteria:

* New York Heart Association class IV congestive heart failure
* Atrial septal defect or atrial septal repair or closure device
* Single occurrence of atrial fibrillation
* Cardioversion or ablation procedure planned within 30 days
* Implanted mechanical valve prosthesis
* Heart transplantation
* Enrolled in another IDE or IND investigation of a cardiovascular device or an investigational drug
* Pregnant or pregnancy is planned during the course of the investigation
* Active infection of any kind
* Severe chronic kidney insufficiency (CrCl< 30 ml/min)
* Terminal illness with life expectancy < 1 yr
* Echocardiographic exclusion criteria
* Left ventricular ejection fraction < 20%
* Intra-cardiac thrombus or dense spontaneous echo contrast as visualized by TEE within 2 days before implant
* Significant mitral valve stenosis (ie, MV <1.5 cm2)
* Complex aortic atheroma with mobile plaque of the descending aorta and/or aortic arch
* Cardiac tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Composite of left atrial appendage (LAA) patency at 45 day evaluated with cardiac computed tomography angiography (CCTA) or the crossover from one device to the other device based on morphological/anatomical considerations during device implantation | 45 days
  Composite endpoint

SECONDARY OUTCOMES:
All cause of death, stroke, systemic or pulmonary embolism and spontaneous myocardial infarction | 48 hours, 45 days, 1 year, 2 years, 3 years, 4 years and 5 years
  Composite endpoint
LAA patency at 45-day and 13-month CCTA in the per protocol and as treated populations | 45 days and 13 months
  LAA patency (arterial and/or venous phase) at 45-day and 13-month CCTA in the per protocol and as treated populations
Cardiovascular death | 48 hours, 45 days, 1 year, 2 years, 3 years, 4 years and 5 years
  Cardiovascular death
Ischemic stroke | 48 hours, 45 days, 1 year, 2 years, 3 years, 4 years and 5 years
  Ischemic stroke
Haemorrhagic stroke | 48 hours, 45 days, 1 year, 2 years, 3 years, 4 years and 5 years
  Haemorrhagic stroke
Bleeding events according to the BARC classification at each follow up | 48 hours, 45 days, 1 year, 2 years, 3 years, 4 years and 5 years
  Bleeding events according to the BARC classification at each follow up
Procedure-related complications | 48 hours, 45 days, 1 year, 2 years, 3 years, 4 years and 5 years
  Procedure-related complications
Rate of patients on (N)OAC at 45 days and 6 months | 45 days and 6 months
  Rate of patients on (N)OAC at 45 days and 6 months
Device thrombosis | 45 days and 13 months
  Device related thrombosis at 45 day TEE/CCTA and 13-month CCTA in the per protocol and as treated populations
Number of device implantation attempts | end of procedure
  Number of device implantation attempts
Total time procedure | end of procedure
  Total time procedure (minutes)
x-ray dose | end of procedure
  x-ray dose (cGy.cm2)
fluoroscopy duration | end of procedure
  fluoroscopy duration (minutes)
amount of contrast used during the procedure | end of procedure
  amount of contrast used during the procedure (ml)
LAA patency | 45 days
  LAA patency at 45 day by TEE in the per protocol and as treated populations

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, Prof, Study Chair — Fondazione Cardiocentro Ticino; Emmanuel Teiger, Prof, Principal Investigator — Hôpital Hôpitaux Universitaires Henri-Mondor; Nicolas Meneveau, Prof, Principal Investigator — Centre Hospitalier Régional Universitaire Hôpital Jean Minjoz; Frederic Anselme, Prof, Principal Investigator — Centre Hospitalier Universitaire Hôpitaux De Rouen; Lorenz Räber, Prof, Study Chair — Inselspital, Bern University Hospital
Locations (8):
- Centre Hospitalier Universitaire de Charleroi, Charleroi, Belgium
- France (4):
  - Centre Hospitalier Régional Universitaire Hôpital Jean Minjoz, Besançon
  - Hopital cardiologique Haut Lévêque CHU de Bordeaux, Bordeaux
  - Hôpital Hôpitaux Universitaires Henri-Mondor, Créteil
  - Centre Hospitalier Universitaire Hôpitaux De Rouen, Rouen
- IRCCS Policlinico S.Donato, Milan, Italy
- Switzerland (2):
  - Bern University Hospital, Bern, Switzerland/Bern
  - Department of Cardiology, Cardiocentro Ticino, Lugano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galea R, De Marco F, Aminian A, Meneveau N, Anselme F, Grani C, Huber AT, Teiger E, Iriart X, Angelillis M, Brugger N, Spirito A, Corpataux N, Franzone A, Vranckx P, Fischer U, Pedrazzini G, Bedogni F, Windecker S, Raber L, Valgimigli M. Design and Rationale of the Swiss-Apero Randomized Clinical Trial: Comparison of Amplatzer Amulet vs Watchman Device in Patients Undergoing Left Atrial Appendage Closure. J Cardiovasc Transl Res. 2021 Oct;14(5):930-940. doi: 10.1007/s12265-020-10095-4. Epub 2021 Apr 21. PMID 33884564
- [Result] Galea R, De Marco F, Meneveau N, Aminian A, Anselme F, Grani C, Huber AT, Teiger E, Iriart X, Babongo Bosombo F, Heg D, Franzone A, Vranckx P, Fischer U, Pedrazzini G, Bedogni F, Raber L, Valgimigli M. Amulet or Watchman Device for Percutaneous Left Atrial Appendage Closure: Primary Results of the SWISS-APERO Randomized Clinical Trial. Circulation. 2022 Mar 8;145(10):724-738. doi: 10.1161/CIRCULATIONAHA.121.057859. Epub 2021 Nov 6. PMID 34747186
- [Derived] Galea R, Perich Krsnik J, Peters AA, De Marco F, Aminian A, Meneveau N, Heg D, Grani C, Anselme F, Franzone A, Vranckx P, Fischer U, Bedogni F, Raber L, Valgimigli M. Incidence and predictors of persistent left atrial appendage patency and its subtypes after percutaneous closure: a pre-specified analysis of the SWISS-APERO trial. Eur Heart J Cardiovasc Imaging. 2025 Oct 30;26(11):1795-1803. doi: 10.1093/ehjci/jeaf232. PMID 40795219
- [Derived] Galea R, De Marco F, Aminian A, Meneveau N, Chalkou K, Anselme F, Grani C, Franzone A, Vranckx P, Fischer U, Valgimigli M, Raber L. 3-Year Clinical Outcomes Comparing the Amulet vs Watchman FLX for Left Atrial Appendage Closure in Patients With Atrial Fibrillation: Results From the SWISS-APERO Randomized Clinical Trial. J Am Coll Cardiol. 2025 Jul 8;86(1):3-14. doi: 10.1016/j.jacc.2025.03.535. PMID 40602941
- [Derived] Galea R, Meneveau N, De Marco F, Aminian A, Heg D, Chalkou K, Grani C, Anselme F, Franzone A, Vranckx P, Fischer U, Bedogni F, Raber L, Valgimigli M. One-Year Outcomes After Amulet or Watchman Device for Percutaneous Left Atrial Appendage Closure: A Prespecified Analysis of the SWISS-APERO Randomized Clinical Trial. Circulation. 2024 Feb 6;149(6):484-486. doi: 10.1161/CIRCULATIONAHA.123.067599. Epub 2023 Oct 24. No abstract available. PMID 37875064
- [Derived] Galea R, Aminian A, Meneveau N, De Marco F, Heg D, Anselme F, Grani C, Huber AT, Teiger E, Iriart X, Franzone A, Vranckx P, Fischer U, Pedrazzini G, Bedogni F, Valgimigli M, Raber L. Impact of Preprocedural Computed Tomography on Left Atrial Appendage Closure Success: A Swiss-Apero Trial Subanalysis. JACC Cardiovasc Interv. 2023 Jun 12;16(11):1332-1343. doi: 10.1016/j.jcin.2023.02.027. Epub 2023 May 3. PMID 37316145

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT03399851/Prot_SAP_000.pdf